CLINICAL TRIAL: NCT07021079
Title: Effects of Focal Muscle Vibration as a Countermeasure Against Hypoactivity-induced Neuromuscular Deconditioning
Brief Title: Muscle Vibration as a Countermeasure Against Hypoactivity-induced
Acronym: NEUROVIB-ULLS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24CH295; 2024-A02769-38 (Other: ID-RCB)
Record Dates: First submitted 2025-03-10; First posted 2025-06-13 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-06

CONDITIONS: Vibration Therapy; Healthy Volunteer Study; Hypoactivity
Keywords: hypoactivity; neuromuscular deconditionning; Vibration
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VIBRATION (Active Comparator): Participants will benefit a local vibration countermeasure program for the knee extensor muscles.
  Interventions: Device: Focal muscle vibration
- CONTROLE (Sham Comparator): the control group WILL not receive this countermeasure.
  Interventions: Device: NO Focal muscle vibration

INTERVENTIONS:
Device: Focal muscle vibration — focal muscle vibration sessions, using small and portable vibrator devices.
  Arms: VIBRATION
Device: NO Focal muscle vibration — The control group will not receive any intervention.
  Arms: CONTROLE

SUMMARY:
Muscle deconditioning, characterized by a loss of muscle mass and strength, is a frequent consequence of prolonged lower limb unloading. Beyond muscle mass loss, reduced neural drive contributes significantly to strength decline, highlighting the need for interventions targeting neuromuscular function during immobilization. Focal muscle vibration (FMV) has shown promise in modulating neuromuscular excitability by activating muscle spindle afferents and inducing cortical adaptations. Chronic use of FMV has been associated with significant strength gains and improved neural command. This makes FMV an effective rehabilitation tool. Its simplicity and non-invasiveness further make it a practical countermeasure.

DETAILED DESCRIPTION:
This study hypothesizes that a 10-day FMV protocol can induce neural adaptations to limit strength loss during unilateral lower limb suspension, offering a novel strategy against neuromuscular function decline.

ELIGIBILITY:
Inclusion Criteria:

* Men and women.
* Aged 18 to 45 years.
* Body Mass Index (BMI) between 20 and 25 kg/m².
* Engaging in at least 1.5 hours per week of physical activity (e.g., brisk walking, running, swimming, cycling).
* Provided informed consent after receiving detailed information about the study.
* Affiliated with or beneficiaries of a social security system

Exclusion Criteria:

* Chronic cardiovascular, neuromuscular, bone, metabolic, and/or inflammatory disorders.
* Personal history and/or risk factors for thrombosis.
* Use of antidepressant medications.
* Use of neuroactive substances likely to alter corticospinal excitability (e.g., hypnotics, antiepileptics, psychotropics, muscle relaxants) during the study.
* Recent bone or ligament trauma within the past 12 months.
* Inability to perform the physical efforts required for the study.
* Recent participation in a sporting competition or intense, unusual physical activity within the past month.
* Corticosteroid treatment within the past 3 months.
* Any skin lesions at the planned vibrator application site.
* Simultaneous participation in another interventional medical study.
* Pregnant or breastfeeding women.
* Individuals unable to understand the purpose and conditions of the study or unable to provide informed consent.
* Individuals deprived of liberty or under guardianship

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Isometric force measurement | Day 1, 7, 14, 28, 33
  Maximal isometric force (% decrease) in knee extension of the immobilized leg will be evaluated

SECONDARY OUTCOMES:
Maximum voluntary force measurement | Day 1, 7, 14, 28, 33
  Maximum voluntary force (Nm) in knee extension, assessed in isometric (for the immobilized leg and also for the contralateral leg), concentric (+60°/s and +180°/s) and eccentric (-60°/s) conditions.
Jumping performance measurement | Day 1, 7, 14, 28, 33
  Jumping performance (height, in cm), assessed in vertical jump tests (Squat Jump and Counter Movement Jump).
Postural balance measurement | Day 1, 7, 14, 28, 33
  Postural balance performance (displacement of center of pressure, in mm), assessed in a unipodal postural balance test performed on a strength platform
Neuromuscular fatigue measurement | Day 1, 7, 14, 28, 33
  Neuromuscular fatigue (decrease in maximum voluntary force (in %), assessed during a fatigue protocol consisting of quadriceps muscle contractions at incremental force levels.
Force-velocity-endurance measurement | Day 1, 7, 14, 28, 33
  Force-velocity-endurance profile, assessed during an effort performed on a cycloergometer at linearly decreasing power values.
Voluntary activation level evaluation | Day 1, 7, 14, 28, 33
  Voluntary activation level (in %), determined by the force increment obtained following stimulation during a maximal voluntary isometric contraction.
Cortico-spinal excitability measurement | Day 1, 7, 14, 28, 33
  Cortico-spinal excitability, assessed by electromyographic responses (motor evoked potentials, in mV) evoked by transcranial magnetic stimulation (TMS).
Spinal excitability evaluation | Day 1, 7,14 , 28, 33
  Spinal excitability (i.e. spinal reflexes, in mV), assessed by recording EMG responses evoked by electrical stimulation of the lumbar vertebrae.
Cortical activation of sensorimotor areas measurement | Day 1, 7, 14, 28, 33
  Cortical activation of sensorimotor areas, assessed by recording the electroencephalographic (EEG) signal during submaximal isometric contractions.
Muscle volume measurement | Day 1, 7, 14, 28, 33
  Muscle volume will be assessed by ultrasound of the thigh muscles (in cm2).
Determination of plasma molecular markers of bone and muscle remodeling | Day 1, 7, 14, 28, 33
  Assessment of blood factors of nerve (BDNF) and muscle remodeling (circulating steroids, insulin, GH, IGF-1, myostatin, activinA, follistatin).
Determination of plasma molecular markers of bone and muscle remodeling | Day 1, 7, 14, 28, 33
  Evaluation of bone remodeling factors by bAP, CTx, P1NP and Trap5b assays
Plasma molecular markers of thrombotic risk evaluation | Day 1, 7, 14, 28, 33
  Plasma molecular markers of thrombotic risk will be assessed by blood sampling followed by assay of HSP47 and D-dimer factors.

CONTACTS AND LOCATIONS:
Overall Officials: LEONARD FEASSON, PHD, Principal Investigator — CENTRE HOSPITALIER UNIVERSITAIRE SAINT-ETIENNE
Locations (1):
- Centre Hospitalier Universitaire, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No